CLINICAL TRIAL: NCT05414097
Title: Finding Barriers and Designing Solutions to Promote Women s Cancer Screening in South Africa
Acronym: FIND
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Other Study IDs: IGHID12101; R21TW011715-01 (NIH)
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Cervical Cancer
Keywords: sequential mixed-methods; HIV; screening
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Growth and Development

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Phase 1: 24 Women - FGDs: Focus groups enrolling HIV-positive, previously screened for cervical cancer; HIV-positive, not previously screened for cervical cancer; HIV-negative, previously screened for cervical cancer; HIV-negative, not previously screened for cervical cancer.
  Interventions: Other: Semi-structured focus group discussions - Women
- Phase 1: 16 Men - FGDs: Focus groups enrolling male partners referred by women previously screened or treated for cervical cancer and by women not previously screened for cervical cancer.
  Interventions: Other: semi-structured focus groups discussions - Men
- Phase 1: 12 Key Stakeholders - IDIs: Stakeholder interviewers with women's groups, women's health providers, laboratory personnel, NGOs, and public health organizations.
  Interventions: Other: In-depth key stakeholders interviews
- Phase 2: 300 women - DCE: Discrete Choice Experiment enrolling women 18 years of age and older.
  Interventions: Other: Discrete Choice Experiment - Women
- Phase 3: 36 Women, women's health providers, and policy makers: Stakeholder groups comprising individuals 18 years and older who participated in Phase 1 will be eligible.
  Interventions: Other: Development and User Pre-testing Workshops

INTERVENTIONS:
Other: Semi-structured focus group discussions - Women — Semi-structured focus group discussions to explore women's experiences with cervical cancer screening and treatment.
  Groups: Phase 1: 24 Women - FGDs
Other: semi-structured focus groups discussions - Men — Semi-structured focus group discussions to explore partner dynamics related to women's ability to access cancer screening.
  Groups: Phase 1: 16 Men - FGDs
Other: In-depth key stakeholders interviews — In-depth interviews to contextualise findings from women and men focus group discussions.
  Groups: Phase 1: 12 Key Stakeholders - IDIs
Other: Discrete Choice Experiment - Women — Discrete Choice Experiment to determine preferences to different cancer screening models.
  Groups: Phase 2: 300 women - DCE
Other: Development and User Pre-testing Workshops — Development and User Pre-testing Workshops to explore acceptability and feasibility of proposed interventions designed using findings from Phases 1 &2.
  Groups: Phase 3: 36 Women, women's health providers, and policy makers

SUMMARY:
The primary aim of the study explore drivers of cervical cancer screening and barriers contributing to low screening coverage among women in South Africa. Secondary aims are determining preferences for cervical cancer prevention services using a discrete choice experiment and developing a multi-level package of interventions that will address barriers to cervical cancer screening and improve engagement in care among women.

DETAILED DESCRIPTION:
Cervical cancer is a leading cause of cancer death among South African women. Despite a comprehensive national cancer control policy, cervical screening coverage is low and attrition during on-ward referrals for diagnostic confirmation and treatment remains common.

This study uses a sequential mixed-methods design:

Phase 1) A qualitative exploratory phase using focus groups and in-depth interviews with women, men, other stakeholders will inform our design and interpretation of quantitative findings from a multi-cohort DCE.

Phase 2) Women will be recruited to participate in the DCE and determine their preferences for cancer screening services.

Phase 3) Design Thinking to co-create an intervention package for cervical cancer screening and enhanced linkage between screening, diagnosis, and treatment will be created.

ELIGIBILITY:
Inclusion Criteria

Focus Groups with HIV-positive Women

1. HIV-positive
2. Women 18 years and older
3. Participants should be willing and able to provide written informed consent

Focus Groups with HIV-negative Women

1. HIV-negative
2. Women 18 years and older
3. Participants should be willing and able to provide written informed consent

Focus Groups with Men

1. Male partners who are 18 years and older
2. Participants should be willing and able to provide written informed consent

In-depth Interviews with Key Stakeholders

1. Healthcare providers working within the public health system and other key stakeholders
2. Individuals 18 years and older
3. Participants should be willing and able to provide written informed consent

Exclusion Criteria:

Focus Groups with HIV-positive Women

1. Women younger than 18 years
2. Unwilling or unable to provide written informed consent

Focus Groups with HIV-negative Women

1. Women younger than 18 years
2. Unwilling or unable to provide written informed consent

Focus Groups with Men

1. Male partners younger than 18 years
2. Participants unwilling or unable to provide written informed consent

In-depth Interviews with Key Stakeholders

1. Providers who do not work in the public health system
2. Individuals younger than 18 years
3. Participants unwilling or unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants for the study will be recruited from both urban and peri-urban settings in Johannesburg, South Africa. The population consists of women who have previously undergone screening/treatment for cervical cancer and those who have not; male partners of these women; and key stakeholders within public health systems.
Sampling Method: Non-Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2022-07-16 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Phase 1: Barriers to cancer screening and engagement | Single visit
  Barriers and enablers will be explored through focus groups and in-depth interviews with women, men, and other stakeholders.

SECONDARY OUTCOMES:
Phase 2: Woman preferences for cancer screening services | Single visit
  Preferences for cancer screening will be determined through the relative importance of the attribute according on how it is scored in the Discrete Choice Experiment.
Phase 3: Acceptability and feasibility of multi-level package of interventions addressing barriers to cancer screening. | Single visit
  Acceptability and feasibility will be measured through development and user pre-testing workshops.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Chibwesha, MD, MSc, Principal Investigator — Department of Obstetrics and Gynecology University of North Carolina at Chapel Hill
Locations (1):
- Clinical HIV Research Unit Temba Lethu Wing Helen Joseph Hospital, Westdene, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: No
Deidentified individual data will however be shared widely. We will make research datasets available to South African investigators who request access and meaningfully involve in-country investigators in all our activities, including the production of research manuscripts and presentations at scientific meetings. All data sharing will abide by rules and/or policies defined by the sponsor, relevant IRBs, U.S. local, state, and federal laws and regulations, as well as South African laws and regulations. Data sharing mechanisms will ensure that the rights and privacy of individuals participating in NIH sponsored research will be protected at all times.

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials